CLINICAL TRIAL: NCT07372742
Title: Clinical Characteristics and Epidemiology of Chronic Critically Ill Patients in China
Status: Recruiting | Type: Observational
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Yi Ji, Professor, West China Hospital
Other Study IDs: 2026-01-12
Record Dates: First submitted 2026-01-19; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Chronic Critically Ill

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to enroll chronic critically ill patients in ICU to investigate the epidemiology of chronic critically ill in China and identify risk factors of poor outcomes among those patients. The main question it aims to answer is:

What is the one year mortality of chronic critically ill patients in China? We conduct semi-structured telephone follow-ups to investigate the long-term outcomes of chronic critically ill patients.

ELIGIBILITY:
Inclusion Criteria:

- Must meet: Age greater than 18 years old; Stay in ICU for 8 days or more.

Meet any of the following criteria:

Tracheotomy; Continuous mechanical ventilation for over 96 hours; Multiple organ failure; Sepsis or severe infection; Severe trauma; Severe brain injury;

Exclusion Criteria:

- Refusing to accept follow-up; Patients who have been lost to follow-up;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a prospective cohort study that will consecutively enroll patients meeting the criteria for Chronic Critical Illness (CCI) from the Intensive Care Units of several hospitals in China over a one-year period starting March 2025.
Sampling Method: Probability Sample
Enrollment: 459 (Estimated)
Dates: Start 2025-03-29 (Actual); Primary Completion 2029-02-01 (Estimated); Study Completion 2029-06-01 (Estimated)

PRIMARY OUTCOMES:
one year mortality | one year
  one year mortality

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital of Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No